CLINICAL TRIAL: NCT07337330
Title: Comparative Study Between Ultrasound Guided External Oblique Intercostal Plane Block and Erector Spinae Block for Postoperative Analgesia in Hepatectomy Incision in Cancer Patients
Brief Title: Ultrasound Guided External Oblique Intercostal Plane Block Versus Erector Spinae Block for Post Hepatectomy Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Asmaa Elsayed Khalil, Lecturer of Anaesthesia, Surgical ICU and Pain Management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AP2509-501-126-203
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pain; Cancer; Hepatectomy; Nerve Block
Keywords: hepatectomy; erector spinae block; external oblique intercostal plane block; liver cancer; ultrasound guided
MeSH Terms: conditions — Cancer Pain; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- External Oblique Intercostal (EOI) Plane Block (Active Comparator): Patient lies supine with their ipsilateral arm abducted. A 12-15 MHz linear transducer will be used. The proceduralist scans the chest wall while at the patient's ipsilateral shoulder. The probe is placed in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle (EOM) is identified at the level of ribs 6 &7 in line with the xiphoid process. To confirm identification of the EOM, the probe is moved caudally following the EOM. At the subcostal level, the ultrasound probe is rotated 90° to see the convergence of the internal oblique & transversus abdominus muscles. The probe is then moved back to the initial identification point. The EOI plane is identified deep to the external oblique and superficial to the 6th & 7th ribs and their associated intercostal muscles. Local anaesthetic is injected subcutaneously & a 16 G Tuohy needle is inserted caudally; the EOI plane is hydrodissected with saline, injecting 20 ml of 0.25% bupivacaine.
  Interventions: Procedure: Ultrasound guided external oblique intercostal (EOI) plane block
- Erector Spinae (ESP) Block (Active Comparator): The patient lies in lateral position, then spinous processes are palpated and marked directly on the skin by a dermographic pencil, and the correctness of the final marking is confirmed by sonographic inspection. A 21G, 50 mm needle isinserted with a cephalad-to-caudal direction into the posterior thoracic wall at the T5 level, to reach the respective transverse process. The proper needle tip positioning ischecked by ultrasound guidance with a 12.5 MHz linear probe (FUJIFILM Sonosite M-Turbo C Ultrasound System) the visualization of a linear fluid spread that distended the fascial plane between the erector spinae muscles group and the transverse process while injecting 2 mL of normal saline solution isconsidered confirmatory. Subsequently, 20 mL of local anaesthetic injected 0.25% bupivacaine
  Interventions: Procedure: Ultrasound guided erector spinae block

INTERVENTIONS:
Procedure: Ultrasound guided external oblique intercostal (EOI) plane block — Patient lies supine with their ipsilateral arm abducted. A 12-15 MHz linear transducer will be used. The proceduralist scans the chest wall while at the patient's ipsilateral shoulder. The probe is placed in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle (EOM) is identified at the level of ribs 6 &7 in line with the xiphoid process. To confirm identification of the EOM, the probe is moved caudally following the EOM. At the subcostal level, the ultrasound probe is rotated 90° to see the convergence of the internal oblique & transversus abdominus muscles. The probe is then moved back to the initial identification point. The EOI plane is identified deep to the external oblique and superficial to the 6th & 7th ribs and their associated intercostal muscles. Local anaesthetic is injected subcutaneously & a 16 G Tuohy needle is inserted caudally; the EOI plane is hydrodissected with saline, injecting 20 ml of 0.25% bupivacaine.
  Arms: External Oblique Intercostal (EOI) Plane Block
Procedure: Ultrasound guided erector spinae block — The patient lies in lateral position, then spinous processes are palpated and marked directly on the skin by a dermographic pencil, and the correctness of the final marking is confirmed by sonographic inspection. A 21G, 50 mm needle isinserted with a cephalad-to-caudal direction into the posterior thoracic wall at the T5 level, to reach the respective transverse process. The proper needle tip positioning ischecked by ultrasound guidance with a 12.5 MHz linear probe (FUJIFILM Sonosite M-Turbo C Ultrasound System) the visualization of a linear fluid spread that distended the fascial plane between the erector spinae muscles group and the transverse process while injecting 2 mL of normal saline solution isconsidered confirmatory. Subsequently, 20 mL of local anaesthetic injected 0.25% bupivacaine
  Arms: Erector Spinae (ESP) Block

SUMMARY:
Management of acute post-operative pain has received keen attention in recent years with considerable concurrent advancement in the field.

The importance of effective pain relief has long been realised, and acute pain services (APS) are operational in majority of the hospitals in the developed world for decades.

Postoperative pain following abdominal surgery if severe enough may cause several side effects as "splinting, hypoventilation, atelectasis, immobility, hypercoagulability, thromboembolic events, vasoconstriction, tachycardia, increased systemic vascular resistance, dysrhythmias and cardiac ischemia in susceptible patients, insomnia, anxiety, feeling of helplessness".

Ultrasound-guided fascial plane blocks have been rapidly incorporated into regional anaesthesia practice in recent years as an alternative to neuraxial techniques and involve injection into a tissue plane to provide analgesia in various anatomic areas.

External oblique intercostal plane block (EOIPB) is a novel block, which has been described as an important modification of the fascial plane blocks that can consistently involve the upper lateral abdominal walls.

The erector spinae plane (ESP) block is a new regional aesthetic technique that can be used to provide analgesia for a variety of surgical procedures or to manage acute or chronic pain. The technique is relatively easy to perform on patients.

The ESPB involves injection of local anaesthetic in the erector spinae fascial plane, superficial to the tip of the transverse process of the vertebra and deep to the erector spinae muscle.

DETAILED DESCRIPTION:
A 20G IV cannula will be inserted. All patients will be premedicated with IV midazolam 0.01-0.02 mg/kg 30 minutes preoperatively. all patients will be monitored continuously using ECG, NIBP, peripheral arterial oxygen saturation and end tidal carbon dioxide throughout the duration of surgery.

Induction of general anaesthesia will be done by propofol 1.5-2 mg/kg, fentanyl 1-2 μg/kg, and atracurium 0.5 mg/kg IV. All patients will receive paracetamol 1 gm by IV drip, ketorolac 30 mg IV drip. Anaesthesia will be maintained by sevoflurane 2%-3% in O2/air mixture with reinjection of atracurium 0.1 mg/kg every 30 minutes. The same procedures will be applied to all patients.

Group 1 - External Oblique Intercostal Block (EOI) Patients positioned in the supine position with their ipsilateral arm abducted. A 12-15 MHz linear transducer (FUJIFILM Sonosite M-Turbo C Ultrasound System) will be used for ultrasonography. With the proceduralist at the patient's ipsilateral shoulder, the chest wall is systematically scanned. Initially the probe is placed in a cephalad to caudad paramedian direction at the anterior axillary line, and the external oblique muscle identified at the level ribs 6 and 7 in line with the xiphoid process. To confirm correct identification of the external oblique muscle, the probe is moved in the caudad direction following the external oblique muscle. At the subcostal level, the ultrasound probe is rotated 90° to see the convergence with the internal oblique and transversus abdominus muscles. The probe is then moved back to the initial identification point for the external oblique muscle. The EOI plane is identified deep to the external oblique muscle and superficial to the sixth and seventh ribs and their associated intercostal muscles. Local anaesthetic is then infiltrated subcutaneously and a 16 G Tuohy needle is inserted cephalad to caudad, and the EOI plane was hydro-dissected with saline,20 ml of local anaesthetic injected (0.25% bupivacaine)(8).

Group 2 - Erector Spinae Block (ESP) The patient in lateral position, then spinous processes were palpated and marked directly on the skin by a dermographic pencil, and the correctness of the final marking was confirmed by sonographic inspection. A 21-gauge, 50 mm needle was inserted with a cephalad-to-caudal direction into the posterior thoracic wall at the T5 level, to reach the respective transverse process.

The proper needle tip positioning was checked by ultrasound guidance with a 12.5 MHz linear probe (FUJIFILM Sonosite M-Turbo C Ultrasound System) the visualization of a linear fluid spread that distended the fascial plane between the erector spinae muscles group and the transverse process while injecting 2 mL of normal saline solution was considered confirmatory.

Subsequently, 20 mL of local anaesthetic injected 0.25% bupivacaine (9).

Intraoperative rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels. Ringer acetate will be infused to replace the fluid deficit, maintenance and losses, and the patients will be mechanically ventilated at appropriate settings that keep end-tidal CO2 at 30- 35 mmHg.

The 1st reading of mean arterial pressure (MAP) and heart rate (HR) will be recorded before induction of general anaesthesia to be defined as a baseline reading while another reading will be noted immediately before surgical incision and at 15-minute intervals intraoperatively.

At the end of surgery residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes.

The patients will be transferred to the post-anaesthesia care unit (PACU) where the Visual Analogue Scale score (VAS), MAP and heart rate will be noted immediately on arrival, and the patients will be observed till fulfilling the criteria of discharge then transferred to the ward where multimodal analgesia will be provided as the following: IV paracetamol 1 g /8 hours and IV ketorolac 30mg/8 hours.

Post-operative rescue analgesia will be provided in the form of IV morphine 0.1 mg per kg if the patient VAS Score ≥ 4. The total amount of morphine given in 24 hours will be recorded for both groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed. VAS, MAP, and heart rate will be noted at 1, 6, 12, and 24 hours postoperatively. Side effects of morphine include: nausea, vomiting, sedation, and respiratory depression (respiratory rate <10/minute), and they will be recorded.

Postoperative nausea and vomiting (PONV) will be rated on a four-point verbal scale; (none =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe =vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients undergoing hepatectomy under general anaesthesia
* Aged 18 years or older
* ASA II & III
* BMI >20kg/m2 and <35kg/m2

Exclusion Criteria:

* History of psychiatric disorders or history of major depression.
* Major medical conditions (heart failure , chronic kidney disease ,patient on dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Pain scores using Visual analogue score | 24 hours after surgery
  Pain scores using Visual analogue score (VAS) (0 mm = no pain to 10mm = worst pain imaginable) at predetermined time intervals (1,6, 12 and 24h) postoperative.

SECONDARY OUTCOMES:
Time of first rescue postoperative analgesia | First 24 hours post-operative
  The total 24-hour morphine consumption will be recorded for every patient post operative.
Total amount of fentanyl consumed intraoperative | Duration of the surgery
  the rescue analgesia will be administered intra-operative by fentanyl IV and the total fentanyl used will be recorded and compared between the groups
Total amount of morphine consumed postoperatively | First 24 hours post-operative
  The total 24-hour morphine consumption will be recorded for every patient post operative.
Post-operative morphine side effects in the post-operative period. | First 24 hours post-operative
  Postoperative nausea and vomiting (PONV), respiratory depression and/or sedation
Changes and stability in Mean Arterial Blood Pressure (MAP) | every 15 minutes during the surgery then at 1, 6, 12 and 24 hours postoperatively
  Change in Mean Arterial Blood Pressure (MAP) in mmHg
Changes and stability in Heart Rate (HR) | every 15 minutes during the surgery then at 1, 6, 12 and 24 hours postoperatively
  Change in heart rate (HR) in beat\min

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mohamed, MD, Principal Investigator — National Cancer Institute Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saad SI, Abd El-Hamid AM, Elbarbary DH, Taher MG. Analgesic Efficacy of Ultrasound-Guided Erector Spinae Plane Block versus Transversus Abdominis Plane Block for Post-Operative Pain Relief in Patients Scheduled for Abdominal Surgeries. Benha medical journal, 2023; 40: 32-48
- [Background] Bonvicini D, Boscolo-Berto R, De Cassai A, Negrello M, Macchi V, Tiberio I, Boscolo A, De Caro R, Porzionato A. Anatomical basis of erector spinae plane block: a dissection and histotopographic pilot study. J Anesth. 2021 Feb;35(1):102-111. doi: 10.1007/s00540-020-02881-w. Epub 2020 Dec 19. PMID 33340344
- [Background] White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. No abstract available. PMID 35249704
- [Background] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545
- [Background] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Background] Clarke HA, Manoo V, Pearsall EA, Goel A, Feinberg A, Weinrib A, Chiu JC, Shah B, Ladak SSJ, Ward S, Srikandarajah S, Brar SS, McLeod RS. Consensus Statement for the Prescription of Pain Medication at Discharge after Elective Adult Surgery. Can J Pain. 2020 Mar 8;4(1):67-85. doi: 10.1080/24740527.2020.1724775. PMID 33987487
- [Background] Jindal S, Sidhu GK, Baryha GK, Singh B, Kumari S, Mahajan R. Comparison of efficacy of thoracic paravertebral block with oblique subcostal transversus abdominis plane block in open cholecystectomy. J Anaesthesiol Clin Pharmacol. 2020 Jul-Sep;36(3):371-376. doi: 10.4103/joacp.JOACP_148_19. Epub 2020 Sep 26. PMID 33487905
- [Background] Afshan G, Khan RI, Ahmed A, Siddiqui AS, Rehman A, Raza SA, Kerai R, Mustafa K. Post-operative pain management modalities employed in clinical trials for adult patients in LMIC; a systematic review. BMC Anesthesiol. 2021 May 25;21(1):160. doi: 10.1186/s12871-021-01375-w. PMID 34034672
- [Background] Dengler KL, Brooks DI, Gruber DD. Multimodal approach to postoperative pain is clinically important. Am J Obstet Gynecol. 2022 Aug;227(2):369. doi: 10.1016/j.ajog.2022.05.004. Epub 2022 May 11. No abstract available. PMID 35562050
- [Background] Linzbach A, Nitschke D, Rothaug J, Komann M, Weinmann C, Schleussner E, Meissner W, Jimenez Cruz J, Schneider U. Peripartal pain perception and pain therapy: introduction and validation of a questionnaire as a quality instrument. Arch Gynecol Obstet. 2022 Jun;305(6):1409-1419. doi: 10.1007/s00404-021-06246-w. Epub 2021 Sep 20. PMID 34542680